CLINICAL TRIAL: NCT05538143
Title: Improving Management of Emergency Department Patients With Undifferentiated Syncope: Prospective Validation of the Canadian Syncope Risk Score
Status: Enrolling by invitation | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 1721270
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive ED syncope/presyncope management tool — This is a data-only, prospective observational cohort study to validate the performance metrics of the Canadian Syncope Risk Score in a diverse population of patients evaluated in community EDs of a U.S. integrated health care system.

SUMMARY:
Among Kaiser Permanente Northern California (KPNC) health plan members, age ≥16 years, with recent syncope and presyncope undergoing emergency department (ED) management with a point-of-care clinical decision support (CDS) tool, how well does the Canadian Syncope Risk Score predict 30-day serious outcomes that were not evident during index ED evaluation?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16y
* Member of Kaiser Permanente Northern California (KPNC) health plan
* Presentation to the ED with an ED diagnosis of recent syncope or presyncope (<24h) without a serious etiology identified during the initial ED diagnostic assessment, that is, patients with unexplained syncope.
* Subjects who meet criteria will be identified electronically within the CDS tool in the electronic health record.

Exclusion Criteria:

* Age <16 years old
* Non-members of KPNC
* Patients with obvious witnessed seizure, prolonged loss of consciousness (>5 minutes), post-traumatic loss of consciousness, and new mental status changes
* Patients requiring hospitalization for traumatic injuries (e.g., syncope leading to motorized vehicle collision), because their outcomes may be related to trauma rather than syncope
* Patients with impaired communication capacity, e.g., intoxication, language barriers, and dementia.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to KPNC emergency departments with eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with arrhythmic and nonarrhythmic serious outcomes | 30 days
  Serious outcomes include those which are arrhythmic (arrhythmias, interventions for arrhythmia, or unknown cause of death) and nonarrhythmic (e.g., myocardial infarction, structural heart disease, pulmonary embolism, or hemorrhage)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Kaiser Permanente Oakland Emergency Department, Oakland, California
  - Kaiser Permanente Richmond Emergency Department, Richmond, California
  - Kaiser Permanente Roseville Emergency Department, Roseville, California
  - Kaiser Permanente South Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente Sacramento Emergency Department, Sacramento, California

IPD SHARING:
Plan to Share IPD: No